CLINICAL TRIAL: NCT06579092
Title: A Phase IIb Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety and Tolerability of AZD5004 in Participants Living With Obesity or Overweight With Comorbidity
Brief Title: Effects of AZD5004 in Adults Who Are Living With Obesity or Overweight With at Least 1 Weight-related Comorbidity
Acronym: VISTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D7260C00001; 2024-513691-18-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Obesity or Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1 (Experimental): Active IMP
  Interventions: Drug: AZD5004
- Arm 2 (Experimental): Active IMP
  Interventions: Drug: AZD5004
- Arm 3 (Experimental): Active IMP
  Interventions: Drug: AZD5004
- Arm 4 (Experimental): Active IMP
  Interventions: Drug: AZD5004
- Arm 5 (Experimental): Active IMP
  Interventions: Drug: AZD5004
- Arm 6 (Placebo Comparator): Matching placebo for each of the 5 active arms
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5004 — AZD5004 film-coated tablet once daily during 36 weeks
  Other Names: Active IMP
  Arms: Arm 1; Arm 2; Arm 3; Arm 4; Arm 5
Drug: Placebo — Placebo matching AZD5004 film-coated tablet once daily during 36 weeks
  Arms: Arm 6

SUMMARY:
A Phase IIb, global, randomized, parallel-group, double-blind, placebo-controlled, multicenter study to assess the efficacy and safety of AZD5004 compared with placebo, given once daily as an oral tablet(s) for 36 weeks, in male and female participants at least 18 years of age who are living with obesity (body mass index [BMI] ≥ 30 kg/m2), or overweight (BMI ≥ 27 kg/m2) who have at least 1 weight-related comorbidity

DETAILED DESCRIPTION:
This is a Phase IIb, global, randomized, parallel-group, double-blind, placebo-controlled, multicenter study to assess the efficacy and safety of 5 doses of AZD5004 compared with placebo, given once daily as an oral tablet or tablets for a duration of 36 weeks, in adults aged 18 years and above, who are living with obesity (BMI ≥ 30 kg/m2), or overweight (BMI ≥ 27 kg/m2) and have at least 1 weight-related comorbidity (Hypertension, Dyslipidemia or hyperlipidemia, CV disease and/or Obstructive sleep apnea). Approximately 304 participants will be randomized in the study. The dual primary endpoints are percent change in body weight from baseline at 26 weeks and the proportion of participants with weight loss ≥ 5% of baseline weight at 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age.
* BMI of (a) ≥ 30 kg/m2, or (b) ≥ 27 kg/m2 and have a current diagnosis of at least 1 of the following weight-related comorbidities (treated or untreated):

  (i) Hypertension (ii) Dyslipidemia or hyperlipidemia (iii) CV disease (iv) Obstructive sleep apnea
* A stable body weight for 3 months prior to Screening (± 5% body weight change).

Exclusion Criteria:

* Have obesity induced by other endocrine disorders, such as Cushing's syndrome or monogenic or syndromic obesity such as Prader-Willi syndrome.
* Has received prescription or non-prescription medication for weight loss within the last 3 months prior to Screening.
* Previous or planned (within study period) bariatric surgery or fitting of a weight loss device (eg, gastric balloon or duodenal barrier).
* History of type 1 diabetes mellitus or type 2 diabetes mellitus.
* Clinically significant inflammatory bowel disease, gastroparesis, severe disease, or surgery affecting the upper GI tract.
* History of acute or chronic pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Percent change in body weight from baseline | 26 weeks
  To determine whether AZD5004 is superior to placebo for weight loss
Achieved Weight Loss ≥ 5% From Baseline | 26 weeks
  To determine whether AZD5004 is superior to placebo on achieving weight loss ≥ 5% from baseline

SECONDARY OUTCOMES:
Percent change in body weight from baseline | 36 weeks
  To determine whether AZD5004 is superior to placebo for weight loss
Achieved weight loss ≥ 5% from baseline | 36 weeks
  To determine whether AZD5004 is superior to placebo on achieving weight loss ≥ 5% from baseline
Absolute change from baseline in body weight | Week 26 and Week 36
  To determine whether AZD5004 is superior to placebo for absolute weight loss
Achieved weight loss ≥ 10% as well as ≥ 15% from baseline | Week 26 and Week 36
  To assess the effect of AZD5004 versus placebo on achieving weight loss ≥ 10% as well as ≥ 15% from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Prof Melanie Davies, MBChB MD, Principal Investigator — Diabetes Research Centre Leicester Diabetes Centre - Bloom University of Leicester
Locations (60):
- United States (30):
  - Research Site, Chandler, Arizona
  - Research Site, Huntington Park, California
  - Research Site, La Mesa, California
  - Research Site, Lincoln, California
  - Research Site, Walnut Creek, California
  - Research Site, Hialeah, Florida
  - Research Site, Orlando, Florida
  - Research Site, Lombard, Illinois
  - Research Site, Valparaiso, Indiana
  - Research Site, West Des Moines, Iowa
  - Research Site, Roslindale, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Chesterfield, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Vestal, New York
  - Research Site, Durham, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Beachwood, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, North Charleston, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Woodway, Texas
  - Research Site, Ogden, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Manassas, Virginia
- Australia (4):
  - Research Site, Heidelberg
  - Research Site, Merewether
  - Research Site, St Albans
  - Research Site, St Leonards
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Surrey, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Guelph, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Terrebonne, Quebec
- Germany (7):
  - Research Site, Bad Oeynhausen
  - Research Site, Berlin
  - Research Site, Hamburg
  - Research Site, Mannheim
  - Research Site, Münster
  - Research Site, Oldenburg
  - Research Site, Sankt Ingbert
- Research Site, Suita-shi, Japan
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (6):
  - Research Site, Blackpool
  - Research Site, Bristol
  - Research Site, Chesterfield
  - Research Site, Leicester
  - Research Site, Rotherham
  - Research Site, Witney

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/